CLINICAL TRIAL: NCT05552352
Title: VRAP-Heart - Virtual Reality Assisted Patient Empowerment for Interventions in Structural Heart Disease - A Randomized-Controlled Multicenter Study
Brief Title: VRAP-Heart - Virtual Reality Assisted Patient Empowerment for Interventions in Structural Heart Disease
Acronym: VRAP-Heart
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VRAP-Heart
Record Dates: First submitted 2022-09-12; First posted 2022-09-23 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Severe Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Two-armed, randomized with controlled parallel groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Patients in the intervention arm receive on the day before the implantation of the artificial aortic valve, a virtual reality assisted information. On the day of the implantation the patients are informed about the process via virtual reality assisted information.
  Interventions: Other: Virtual Reality assisted information
- Control Arm (No Intervention): Patients in the control arm receive no virtual reality assisted information.

INTERVENTIONS:
Other: Virtual Reality assisted information — Patients in the intervention group receive a VR instructional application in the patient's room the day before TAVI implantation and in the operational suite during TAVI implantation the next day. In this application, the patient is guided through different VR parts that repeat the indication, the procedure, the localities and the post-interventional phase of the implantation with the corresponding safety instructions.
  Arms: Intervention Arm

SUMMARY:
This prospective, randomized-controlled multicenter study investigates whether virtual reality-assisted patient education in patients undergoing transfemoral transcatheter aortic valve implantation (TAVI) can improve patient understanding and simulative orientation, thereby reducing postinterventional complications, resulting in significantly shorter length of stay.

DETAILED DESCRIPTION:
This prospective, randomized-controlled multicenter study investigates whether VR-assisted patient education in patients undergoing transfemoral transcatheter aortic valve implantation (TAVI) can improve patient understanding and simulative orientation, thereby reducing postinterventional complications, resulting in significantly shorter length of stay. Disorientation, anxiety, and pain can lead to the development of delirium and, through complications, to prolonged hospital stays during elective procedures. Virtual reality can combine different learning modalities (auditory, visual, written, haptic) and improve patient understanding of the procedure through educational interventions. More detailed knowledge of the environment, the players, the procedure, and safety aspects will reduce anxiety and stress before and during the procedure and reduce complications during post-interventional care. As a result, length of stay should be reduced.

ELIGIBILITY:
Inclusion Criteria:

* High-grade aortic valve stenosis
* Indication for elective transfemoral transcatheter aortic valve implantation under analgesia (TAVI)
* Existing heart center decision
* Age ≥ 18 years
* Signed informed consent form

Exclusion Criteria:

* Surgery planned under general anesthesia
* Language barrier, defined as insufficient language proficiency at the discretion of the investigator to understand the purpose of the trial and follow the VR application.
* Severe hearing impairment, preventing the patient from understanding the sound of the VR goggles, tested with the VR goggles fitted without using the VRAP-Heart software
* Severe visual impairment that prevents viewing of the VR modules if it is not possible to use existing visual corrections (contact lenses, glasses) together with the VR glasses in the event of defective vision, tested with the VR goggles fitted without using the VRAP-Heart software
* Moderately severe or severe dementia syndrome noted in the medical history or identified during the informed consent discussion
* Known seizure disorder (epilepsy)
* Positive pregnancy test on inclusion and/or pregnancy is present
* Court ordered placement in an institution
* Any psychosocial condition that makes compliance with the protocol unlikely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay in days | from start of hospitalizations until hospital leave up until day 360
  Primary endpoint is the mean hospital stay in each group in days.

SECONDARY OUTCOMES:
Mental state on the day before the procedure as assessed by visual analog scale | 1 day before procedure
  Anxiety and psychological stress are common before elective procedures such as TAVI. Both are considered triggers and amplifiers of delirium. Patients are asked to quantify their anxiety before the procedure using a visual analog scale ranging from 1 to 10.
Mental state on the day before the procedure as assessed by State-Trait-Anxiety-Inventory questionnaire | 1 day before procedure
  Anxiety and psychological stress are common before elective procedures such as TAVI. Both are considered triggers and amplifiers of delirium. Patients are asked to quantify their anxiety before the procedure using State-Trait-Anxiety-Inventory with minimum outcome 10 and maximum outcome 80. Lesser outcome means more anxiety.
Mental state on the day before the procedure as assessed by Hospital Anxiety and Depression Scale German Version questionnaire | 1 day before procedure
  Anxiety and psychological stress are common before elective procedures such as TAVI. Both are considered triggers and amplifiers of delirium. Patients are asked to quantify their anxiety before the procedure using Hospital Anxiety and Depression Scale German Version questionnaire. Anxiety scale in the questionnaire has values from 0 to 21 and Depression scale has values from 0 to 21. Lesser values denote less anxiety or depression.
Anxiety during the procedure as assessed by visual analog scale | during procedure
  Anxiety and psychological stress are common during elective procedures such as TAVI. Both are considered triggers and amplifiers of delirium. Patients are asked to quantify their anxiety before the procedure using a visual analog scale ranging from 1 to 10.
Anxiety during the procedure as assessed by State-Trait-Anxiety-Inventory questionnaire | during procedure
  Anxiety and psychological stress are common during elective procedures such as TAVI. Both are considered triggers and amplifiers of delirium. Patients are asked to quantify their anxiety before the procedure using State-Trait-Anxiety-Inventory with minimum outcome 10 and maximum outcome 80. Lesser outcome means more anxiety.
Pain during the procedure | during procedure
  Pain can occur despite analgesia during an elective procedure such as TAVI. Pain is considered a trigger and amplifier of delirium. Patients are asked to quantify their pain on a visual analog scale during the procedure (time point: procedure performed but still in the hybrid operating room). Here, 0 corresponds to no pain and 10 to the maximum imaginable pain.
Anxiety/stress before, during, and after surgery (measured as serum cortisol) | on the 1 day before, during and on day 1-3 after procedure
  Anxiety and psychological stress are common before and during elective procedures such as TAVI. Both are considered triggers and amplifiers of delirium. Patients will have routine blood samples taken before, during, and after the procedure. From these, the parameter cortisol in serum is additionally determined optionally in the context of this study. Serum cortisol is an established parameter to quantify anxiety and stress, especially intraindividually.
Anxiety / stress before, during and after the procedure (amylase and cortisol in saliva). | on the 1 day before, during and on day 1-3 after procedure
  Patients will have saliva samples taken before, during and after the procedure. From these, the parameters cortisol and alpha-amylase are additionally determined on an optional basis within the scope of this study. Both parameters are considered established to quantify anxiety and stress especially intraindividually.
Knowledge test after informed consent | 1 day before procedure after informed consent
  In order to test to what extent the addition of a combination of different learning modalities (acoustic, visual, written, haptic) implemented in virtual reality to the medico-legal informed consent is superior to the standard informed consent, a survey is conducted after the informed consent.
Major bleeding and minor bleeding during hospitalization. | at hospital leave up to 360 days after procedure
  Bleeding is a typical complication after cardio-vascular interventional procedures. Unawareness, disorientation, falls, and delirium favor the occurrence of bleeding. After hospital discharge, the occurrence of bleeding is recorded according to Valve Academic Research Consortium-2 consensus document (VARC), which is based on the bleeding academic research consortium (BARC) classification.
Survival / rehospitalization at 6 and 12 months | after 6 and 12 months after hospital leave
  After 6 and 12 months patients are contacted and information is gathered about survival of the patients and possible rehospitalization events.
Maximum length of hospital stay, in days | at hospital leave up to 360 days after procedure
  In addition to the mean hospital stay in days, a maximum hospital stay is also calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Jung, Prof MD PhD, Principal Investigator — Heinrich-Heine University, Duesseldorf
Locations (2):
- Germany (2):
  - Universitätsklinikum Düsseldorf, Klinik für Kardiologie, Pneumologie & Angiologie, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Köln, Klinik III für Innere Medizin, Herzzentrum, Kerpener Straße 62, Cologne

IPD SHARING:
Plan to Share IPD: No